CLINICAL TRIAL: NCT06777953
Title: Comparative Efficacy of Popliteal Sciatic Nerve and Lumbar Sacral Erector Spinae Plane Blocks for Postoperative Analgesia in Tibia Fractures: a Retrospective Cohort Study
Brief Title: Regional Anesthesia for Lower Extremity Surgery
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HEA-AAR-MK-03
Record Dates: First submitted 2025-01-04; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Erector Spinae Plane Block; Lower Extremity Surgery; Sciatic Nerve Block
Keywords: sacral erector spinae plane block; lower extremity surgery; lumbar erector spinae plane block; sciatic nerve block
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Lidocaine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Erector Spinae Plane Block Group: Patients who underwent spinal anesthesia due to tibial fracture will be identified from their follow-up files. Among these patients, those who underwent erector spinae plane block with 20 ml of 0.5% bupivacaine and 5 ml of 1% lidocaine at the sacral level and 20 ml of 0.5% bupivacaine and 5 ml of 1% lidocaine at the L3 level while sitting under ultrasound guidance for postoperative analgesia will constitute this group.
  Interventions: Other: Erector Spinae (ESP) Block with Lidocaine/Bupivacaine
- Sciatic Nerve Plane Block Group: Patients who underwent spinal anesthesia due to tibial fracture will be identified from their follow-up files. Among these patients, those who underwent popliteal sciatic nerve block with 30 ml of 0.5% bupivacaine while supine position under ultrasound guidance for postoperative analgesia will constitute this group.
  Interventions: Other: Popliteal Sciatic Nerve Block

INTERVENTIONS:
Other: Erector Spinae (ESP) Block with Lidocaine/Bupivacaine — This study is to retrospectively compare the analgesic efficacy and impact on postoperative recovery of popliteal sciatic nerve blocks and Lumbar-Sacral Erector Spinae Plane blocks administered for postoperative pain management in tibial fractures.
  Groups: Erector Spinae Plane Block Group
Other: Popliteal Sciatic Nerve Block — This study is to retrospectively compare the analgesic efficacy and impact on postoperative recovery of popliteal sciatic nerve blocks and Lumbar-Sacral Erector Spinae Plane blocks administered for postoperative pain management in tibial fractures.
  Groups: Sciatic Nerve Plane Block Group

SUMMARY:
In this study, patients who underwent osteosynthesis with plate via standard anterolateral incision due to proximal tibia fracture in the orthopedic clinic within the last year; those who underwent perioperative anesthesia with spinal block, those who underwent postoperative analgesia with Ultrasound-guided popliteal sciatic nerve block, lumbar-sacral Erector Spine plane block combinations in the recovery unit will be identified and their files will be scanned retrospectively. Gender, surgical duration, postoperative block, pre-post block pain levels will be reviewed via Visual Analog Scale scoring, postoperative analgesics consumed and their amounts, Bromage scale, mobilization times, block-related complications, satisfaction levels will be determined and these two groups of patients who underwent block will be compared in terms of analgesia, complications, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* Patients undergoing spinal anesthesia
* Patients undergoing postoperative erector spinae plane block
* Patients undergoing postoperative sciatic nerve block

Exclusion Criteria:

* Pregnant patients
* Patients who cannot be contacted
* Patients who have undergone perioperative general anesthesia
* Patients with a history of cerebrovascular disease
* Patients with data loss
* Patients who did not receive consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proximal tibial fractures who underwent surgery within the past year at the orthopedic clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Postoperative Analgesia | 24 hours
  Postoperative analgesia will be assessed by Visual Analog Scale Score and postoperative analgesic consumption. The visual analog scale is a numerical assessment ranging from 0 to 10. A score of 0 is considered as no pain, a score of 5 is considered as moderate pain, and a score of 10 is considered as unbearable pain. Rescue intravenous analgesic treatment is applied to scores of 4 and above.

SECONDARY OUTCOMES:
Block related complication | 24 hours
  Patients will be evaluated with Bromage Scale and mobilization times.The bromage scale is a numerical assessment ranging from 0 to 3. A score of 0 is No motor block, a score of 1 is Inability to raise extended leg; able to move knees and feet no pain, a score of 2 is Inability to raise extended leg and move knee; able to move feet, a score of 3 is Complete block of motor limb.It will also be checked when the patients can walk after the motor block has passed.

CONTACTS AND LOCATIONS:
Overall Officials: Munevver Kayhan, Medical Doctor, Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No